CLINICAL TRIAL: NCT03918447
Title: A Phase 3 Trial of the Efficacy and Safety of Bardoxolone Methyl in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: A Trial of Bardoxolone Methyl in Patients With ADPKD - FALCON
Acronym: FALCON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinuation of all bardoxolone chronic kidney disease programs
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-1808
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Autosomal Dominant Polycystic Kidney; ADPKD
Keywords: Bardoxolone Methyl; RTA 402; Autosomal Dominant Polycystic Kidney Disease; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Maximum bardoxolone methyl dose of 20 mg (Experimental): Patients randomized to receive bardoxolone methyl with a baseline ACR less than or equal to 300 mg/g will be titrated to a maximum dose of 20 mg. Patients will begin once-daily dosing with bardoxolone methyl capsules at 5 mg and will dose escalate to 10 mg at Week 2 and 20 mg at Week 4.
  Patients will continue to receive study drug through Week 100, and will not receive study drug during a 12-week off-treatment period between Weeks 100 and 112.
  Interventions: Drug: Bardoxolone methyl oral capsule
- Maximum bardoxolone methyl dose 30 mg (Experimental): Patients randomized to receive bardoxolone methyl with a baseline ACR greater than 300 mg/g will be titrated to a maximum dose of 30 mg. Patients will begin once-daily dosing with bardoxolone methyl capsules at 5 mg and will dose escalate to 10 mg at Week 2, 20 mg at Week 4 and 30 mg at Week 6.
  Patients will continue to receive study drug through Week 100, and will not receive study drug during a 12-week off-treatment period between Weeks 100 and 112.
  Interventions: Drug: Bardoxolone methyl oral capsule
- Placebo (Placebo Comparator): Patients randomized to placebo will remain on placebo capsules throughout the study, undergoing sham titration.
  Patients will continue to receive placebo capsules through Week 100, and will not receive capsules during a 12-week off-treatment period between Weeks 100 and 112.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Bardoxolone methyl oral capsule — Bardoxolone methyl capsules dose escalated from 5 mg to a maximum of 20 or 30 mg, depending on baseline proteinuria status.
  Other Names: RTA 402
  Arms: Maximum bardoxolone methyl dose 30 mg; Maximum bardoxolone methyl dose of 20 mg
Drug: Placebo oral capsule — Capsule containing an inert placebo
  Arms: Placebo

SUMMARY:
This international, multi-center, randomized, double-blind, placebo-controlled Phase 3 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with ADPKD. Approximately 850 patients will be enrolled.

DETAILED DESCRIPTION:
This international, multi-center, randomized, double-blind, placebo-controlled Phase 3 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with ADPKD.

Patients will be randomized 1:1 to either bardoxolone methyl or placebo. Patients receiving bardoxolone methyl will start with once-daily dosing at 5 mg and will dose-escalate to 10 mg at Week 2, to 20 mg at Week 4, and then to 30 mg at Week 6 (only if baseline ACR >300 mg/g) unless contraindicated clinically and approved by the medical monitor. Dose de-escalation is permitted during the study if indicated clinically, and subsequent dose re-escalation is also permitted to meet the dosing objective of the highest tolerated dose.

All patients in the study will follow the same visit and assessment schedule. Patients will continue to receive study drug or placebo through Week 100 and will not receive study drug or placebo during a 12-week off-treatment period between Weeks 100 and 112.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 ≤ age ≤ 70 upon study consent;
* Diagnosis of ADPKD by modified Pei-Ravine criteria (for adults 18≤ age ≤70 years): 1) at least 3 cysts per kidney by sonography or at least 5 cysts by CT or MRI with family history of ADPKD or 2) at least 10 cysts per kidney by any radiologic method and exclusion of other cystic kidney diseases if without family history;
* Screening eGFR (average of Screen A and Screen B eGFR values) ≥ 30 to≤ 90 mL/min/1.73 m2 (12 to 55 years) or ≥ 30 to ≤ 44 mL/min/1.73 m2 (56 to 70 years):

  1) Patients with either screening eGFR ≥ 60 to ≤ 90 mL/min/1.73 m2 or age 56 to 70 years, must have evidence of ADPKD progression (i.e., eGFR decline of ≥ 2.0 mL/min/1.73 m2 per year, based on historical eGFR data and medical monitor discretion); 2)The two eGFR values collected at Screen A and Screen B visits used to determine eligibility must have a percent difference ≤ 25%;
* Albumin to creatinine ratio (ACR) ≤ 2500 mg/g at Screen B visit;
* Systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg at Screen A or B visit after a period of rest.

Exclusion Criteria:

* History of administration of polycystic kidney disease-modifying agents (somatostatin analogues) within 2 months prior to the Screen A visit;
* B-type natriuretic peptide (BNP) level > 200 pg/mL at Screen A visit;
* Uncontrolled diabetes (HbA1c > 11.0%) at Screen A visit;
* Serum albumin < 3 g/dL at Screen A visit;
* History of intracranial aneurysms;
* Kidney or any other solid organ transplant recipient or a planned transplant during the study;
* Acute dialysis or acute kidney injury within 12 weeks prior to Screen A visit or during Screening;
* History of clinically significant left-sided heart disease and/or clinically significant cardiac disease;
* Systolic BP < 90 mm Hg at Screen A visit after a period of rest;
* BMI < 18.5 kg/m2 at the Screen A visit;
* History of malignancy within 5 years prior to Screen A visit, with the exception of localized skin or cervical carcinomas;
* Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to randomization or anticipated need for immunosuppression during the study;
* Untreated or uncontrolled active bacterial, fungal, or viral infection;
* Participation in other interventional clinical studies within 30 days prior to Day 1;
* Unwilling to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential) during Screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested;
* Women who are pregnant or breastfeeding;
* Concomitant use of tolvaptan is excluded. Patients previously treated with tolvaptan must have discontinued drug for at least 2 months prior to Screen A visit

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (136):
- United States (82):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Nephrology Associates PC, Homewood, Alabama
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - AKDHC, Glendale, Arizona
  - Aventiv Research, Inc, Mesa, Arizona
  - University of Arizona, Tucson, Arizona
  - Rancho Research Institute, Downey, California
  - California Institute Renal Research, La Mesa, California
  - University of California, Los Angeles, Los Angeles, California
  - Keck USC/LAC, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Stanford University, Palo Alto, California
  - Apex Research of Riverside, Riverside, California
  - University of California San Francisco, San Francisco, California
  - Western Nephrology, Arvada, Colorado
  - University of Colorado Anschutz Medical Center, Aurora, Colorado
  - Kidney Associates of Colorado, Denver, Colorado
  - Denver Nephrologist, PC, Denver, Colorado
  - Western Nephrology and Mineral Bone Disease, PC, Westminster, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Pro-Care Research Center, Corp., Miami Gardens, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Innovation Medical Research Center, Inc, Palmetto Bay, Florida
  - Volunteer Medical Research, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Florida Premier Research Institute, LLC, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Nephrology, LLC, Lawrenceville, Georgia
  - Boise Kidney & Hypertension, PLLC, Caldwell, Idaho
  - Boise Kidney & Hypertension, PLLC, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Ascension Via Christi Research, Wichita, Kansas
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - The Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - KidneyCare and Tranplant Services of New England, Springfield, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - Paragon Health PC d/b/a Nephrology Center PC, Kalamazoo, Michigan
  - Michigan Kidney Consultants, Pontiac, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - KSOSN, Las Vegas, Nevada
  - Nephrology Associates, P.C., Flushing, New York
  - Division of Kidney Diseases and Hypertension, Great Neck, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - North Carolina Nephrology, P.A. 2nd Floor, Raleigh, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Nephrology Associates, P.C., Nashville, Tennessee
  - TTUHSC, Amarillo, Texas
  - Arlington Nephrology, PA, Arlington, Texas
  - Research Management, Inc., Austin, Texas
  - Liberty Research Center, Dallas, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - Davita Clinical Research, El Paso, Texas
  - DaVita Med Center, Houston, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Milwaukee Nephrologists, SC, Wauwatosa, Wisconsin
- Australia (10):
  - Renal Research, Gosford, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Melbourne Health, Parkville, Victoria
  - Melbourne Renal Research Group, Reservoir, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (4):
  - Nephrology, Cliniques U St-Luc, Brussels
  - Universitair Ziekenhuis Brussel (VUB), Brussels
  - University Hospitals Leuven, Dept. of Nephrology, Dialysis and Renal Transplantation, Leuven
  - Chu Liege, Liège
- Czechia (3):
  - FN Brno, Brno
  - Nephrology Dept., General Teaching Hospital, Prague
  - IKEM, Prague
- France (5):
  - University Hospital La Cavale Blanche, Brest
  - Chu Grenoble Alpes, Grenoble
  - Hospital Henri-Mondor AP-HP, Le Kremlin-Bicêtre
  - CHU de Nantes, Nantes
  - Hopital Necker, Universite Paris Descartes, Paris
- Germany (3):
  - Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der TU München, München
- Italy (4):
  - Renal Division, ASST Santi Paolo e Carlo, Milan
  - Università di Modena e Reggio Emilia, Modena
  - ICS Maugeri SpA SB, Pavia
  - Fondazione Policlinico Gemelli, Roma
- Japan (10):
  - Hokkaido University Hospital, Hokkaido
  - Toranomon Hospital Kajigaya, Kanagawa
  - Japan Community Healthcare Organization Sendai Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Toranomon Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
- Spain (11):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Del Mar, Barcelona
  - Fundacio Puigvert, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Getafe, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Dr Peset, Valencia
- United Kingdom (4):
  - North Bristol NHS Trust, Bristol
  - Manchester University NHS Foundation Trust, Manchester
  - Nottingham University Hospitals, Nottingham
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in the United States, Australia, Belgium, Czech Republic, France, Germany, Italy, Japan, Spain, and United Kingdom beginning on 29 May 2019. The study completion date was 8 August 2023.
Pre-assignment Details: A total of 667 participants were enrolled and randomized 1:1 to receive either bardoxolone methyl or placebo during the treatment period (up to Week 100) and continued to be assessed in the off-treatment period for 12 weeks (up to Week 112).
Groups:
- Bardoxolone Methyl: During the treatment period, the participants received bardoxolone methyl capsules, once daily (QD) at a starting dose of 5 milligrams (mg), followed by dose-escalation to 10 mg at Week 2, and to 20 mg at Week 4. If the eligibility urine albumin to creatinine ratio (UACR) was >300 milligrams per gram (mg/g), the dose was increased to 30 mg starting from Week 6 until Week 100. Participants continued to be assessed during the off-treatment period up to Week 112.
- Placebo: During the treatment period, participants received bardoxolone methyl matching-placebo capsules, orally, QD up to Week 100, with sham titration to maintain the blinding. Participants did not receive a bardoxolone methyl matching placebo capsule during the off-treatment period between Weeks 100 and 112.
Period: Overall Study
Arm/Group | Bardoxolone Methyl | Placebo
Started | 334 | 333
Safety Analysis Set (Participants who received 1 dose of bardoxolone methyl were classified in the bardoxolone methyl group. Participants who received at least 1 dose of placebo and no dose of bardoxolone methyl were classified in the placebo group.) | 335 | 331
Completed | 106 | 112
Not Completed | 228 | 221
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 13 | 6
Not completed — Withdrawal by Subject | 19 | 17
Not completed — Study Terminated by Sponsor | 195 | 197
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all enrolled participants categorized by their randomized treatment group (whether or not they received study drug).
Groups:
- Bardoxolone Methyl: During the treatment period, the participants received bardoxolone methyl capsules, QD at a starting dose of 5 mg, followed by dose-escalation to 10 mg at Week 2, and to 20 mg at Week 4. If the eligibility UACR was >300 mg/g, the dose was increased to 30 mg starting from Week 6 until Week 100. Participants continued to be assessed during the off-treatment period up to Week 112.
- Total: Total of all reporting groups
Arm/Group | Bardoxolone Methyl | Placebo | Total
Number analyzed (Participants) | 334 | 333 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.46) | 48.3 (9.58) | 48.4 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 173 | 361
  Male | 146 | 160 | 306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 35 | 64
  Not Hispanic or Latino | 305 | 298 | 603
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 1 | 2
  Race: Asian | 34 | 45 | 79
  Race: Black or African American | 23 | 18 | 41
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: White | 269 | 261 | 530
  Race: Other | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Off-treatment Period: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 108
Description: Estimated Glomerular filtration rate (eGFR) is a measure of kidney function assessed through blood/serum. eGFR was measured in milliliters per minute per 1.73 meters square (mL/min/1.73 m^2). Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function. Negative change from baseline in eGFR indicates worsened kidney function.
Time Frame: Baseline, Week 108
Population: ITT population included all enrolled participants categorized by their randomized treatment group (whether or not they received study drug). 'Overall number of participants analyzed' indicates the number of participants with data available for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Bardoxolone Methyl | Placebo
Number analyzed (Participants) | 70 | 79
mL/min/1.73 m^2 | -4.59 (0.817) | -5.56 (0.769)
Statistical Analysis 1: Comparison: Bardoxolone Methyl vs Placebo; ANCOVA model with baseline eGFR as a covariate, and treatment group as fixed effects; Test type: Superiority; p = 0.3886, ANCOVA; Least Square Means Difference = 0.97, 95% CI 2-sided [-1.25 to 3.19], Standard Error of Mean 1.122

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: AE:any untoward medical occurrence in a participant regardless of its causal relationship to study drug.AE can be any unfavorable & unintended sign,symptom/disease temporally associated with use of study drug,whether considered to be study-drug related/not.This includes clinically significant abnormal laboratory test result,any newly occurring events/previous conditions that have increased in severity/frequency since administration of study drug. SAE:any AE that at any dose results in death,life-threatening,requires hospitalization/prolongation of existing hospitalisation,substantial disruption of ability to conduct normal life functions,congenital anomaly or is an important medical event. AEs & SAEs that occurred during treatment and within 30 days after last dose were considered TE.
Time Frame: From first dose of the study drug up to end of follow-up (up to Week 112)
Population: Safety population included all enrolled participants who had received at least 1 dose of study drug. Participants who received 1 dose of bardoxolone methyl were classified in the bardoxolone methyl group. Participants who received at least 1 dose of placebo and no dose of bardoxolone methyl were classified in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Bardoxolone Methyl | Placebo
Number analyzed (Participants) | 335 | 331
Participants
  TEAEs | 314 | 296
  Serious TEAEs | 38 | 26

3. Secondary Outcome: Treatment Period: Change From Baseline in eGFR at Week 100
Description: eGFR is a measure of kidney function assessed through blood/serum. eGFR was measured in mL/min/1.73 m^2. Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function. A negative change from baseline in eGFR indicates worsened kidney function.
Time Frame: Baseline, Week 100
Population: ITT included all enrolled participants categorized by their randomized treatment group (whether or not they received study drug). 'Overall number of participants analyzed' indicates the number of participants with an eGFR assessment at Week 100.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Bardoxolone Methyl | Placebo
Number analyzed (Participants) | 168 | 167
mL/min/1.73 m^2 | 1.31 (0.550) | -6.64 (0.549)
Statistical Analysis 1: Comparison: Bardoxolone Methyl vs Placebo; Mixed model repeated measure (MMRM) model used baseline eGFR as a covariate, and the following fixed factors: treatment group, time (Week 1 to 100, excluding Week 52), and the interaction between treatment and time. Within-participant errors are modeled using an unstructured covariance matrix; Test type: Superiority; p < 0.0001, MMRM; Least Square Means Difference = 7.94, 95% CI 2-sided [6.41 to 9.47], Standard Error of Mean 0.777

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to end of follow-up (up to Week 112)
Description: Safety population included all enrolled participants who had received at least 1 dose of study drug. Participants who received 1 dose of bardoxolone methyl were classified in the bardoxolone methyl group. Participants who received at least 1 dose of placebo and no dose of bardoxolone methyl were classified in the placebo group.
Arm/Group | Bardoxolone Methyl | Placebo
All-Cause Mortality (participants affected / at risk) | 1/335 | 0/331
Serious Adverse Events (participants affected / at risk) | 38/335 | 26/331
Other Adverse Events (participants affected / at risk) | 299/335 | 255/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl (N=335) | Placebo (N=331)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic cyst (Blood and lymphatic system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 2 | 0
Macular degeneration (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Cyst rupture (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 2
Renal cyst infection (Infections and infestations) | 2 | 2
Pneumonia viral (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Corona virus infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Colon injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Renal cyst ruptured (Renal and urinary disorders) | 3 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl (N=335) | Placebo (N=331)
Nausea (Gastrointestinal disorders) | 49 | 40
Constipation (Gastrointestinal disorders) | 38 | 16
Diarrhoea (Gastrointestinal disorders) | 35 | 31
Abdominal pain (Gastrointestinal disorders) | 32 | 21
Vomiting (Gastrointestinal disorders) | 23 | 9
Abdominal distension (Gastrointestinal disorders) | 22 | 9
Fatigue (General disorders) | 47 | 29
Oedema peripheral (General disorders) | 27 | 35
Pyrexia (General disorders) | 22 | 19
Corona virus infection (Infections and infestations) | 76 | 89
Nasopharyngitis (Infections and infestations) | 39 | 31
Upper respiratory tract infection (Infections and infestations) | 26 | 13
Urinary tract infection (Infections and infestations) | 24 | 21
Alanine aminotransferase increased (Investigations) | 76 | 3
Aspartate aminotransferase increased (Investigations) | 47 | 4
Hepatic enzyme increased (Investigations) | 46 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 32 | 23
Brain natriuretic peptide increased (Investigations) | 31 | 16
Weight decreased (Investigations) | 28 | 4
Gamma-glutamyltransferase increased (Investigations) | 24 | 3
Decreased appetite (Metabolism and nutrition disorders) | 26 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 164 | 53
Flank pain (Musculoskeletal and connective tissue disorders) | 43 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 12
Headache (Nervous system disorders) | 55 | 41
Dizziness (Nervous system disorders) | 25 | 13
Renal pain (Renal and urinary disorders) | 12 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 9
Hypertension (Vascular disorders) | 25 | 34

LIMITATIONS AND CAVEATS:
Due to discontinuation of all bardoxolone chronic kidney disease programs, study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03918447/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03918447/SAP_003.pdf